CLINICAL TRIAL: NCT00760552
Title: Trial of Low And High Intensity Strategies to Maintain Blood Pressure Control
Brief Title: Trial of Low and High Intensity Strategies to Maintain BP Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-145
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
Keywords: Hypertension; Adherence; Pharmacist; Interdisciplinary; Randomized Controlled; Primary Care
MeSH Terms: conditions — Hypertension | interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): VA patients with uncontrolled HTN.
  Interventions: Other: High Intensity Intervention; Other: All- 6 month pharmacist intervention
- Arm 2 (Active Comparator): VA patients with uncontrolled HTN.
  Interventions: Other: Low Intensity Intervention; Other: All- 6 month pharmacist intervention

INTERVENTIONS:
Other: High Intensity Intervention — High Intensity patients will be seen by the pharmacist at 3-6 month intervals, depending upon if patient is at goal BP. During these visits, the pharmacist will: 1) review barriers to BP control; 2) assess progress toward overcoming such barriers; 3) determine adherence; and 4) assess potential side effects. If the BP is at goal, the patient will be given encouragement and told to continue the regimen. If the BP is not at goal, the pharmacist will develop a new treatment strategy. If the treatment changes were in the plan negotiated with the physician, the PCP will simply be informed. If new changes are recommended, the pharmacist will develop a new treatment plan and review it with the PCP.
  Arms: Arm 1
Other: Low Intensity Intervention — Low intensity group will receive management by their PCP and a 3-part intervention that was effective in a recent VA study. This one-time intervention will occur 3 months after completion of the initial 6-month pharmacist intervention and will include: Provider education including an email message to re-evaluate the specific patient's BP regimen and a web link to the VA/JNC-7 hypertension guidelines. 1-time patient-specific computerized alert reminding the PCP of the goal BP, values of the patient's last 3 BP assessments, & possible options for medication changes if BP does not remain at goal. Patient education including a personalized letter with information on strategies to improve BP control, including medication adherence, Dietary Approaches to Stop Hypertension (DASH) diet/exercise. The letter will note that many patients require more than one medication and will provide a link to the VA patient education web library and American Heart Association (AHA) site.
  Arms: Arm 2
Other: All- 6 month pharmacist intervention — All patients will receive the initial 6-month pharmacist intervention. The intervention: 1) co-management of HTN by pharmacists can improve BP control; and 2) active follow-up is needed to reinforce progress and proactively identify and resolve problems. The intervention will include structured visits at baseline 1, 2, 4, and 6 months after baseline and telephone calls at 2 weeks and between the visits. At baseline, the pharmacist will review the computerized patient record system (CPRS) medical record and perform a structured interview, including: a detailed medication history of all prescription and non-prescription therapies; an assessment of patient knowledge of all meds, the purpose of each med, medication dosages and timing, and potential side effects; potential contraindications to specific medications; and expectations for future dosage changes and of the need for future monitoring potential barriers to BP control.

SUMMARY:
The long-range goal of this research is to advance understanding of long-term blood pressure (BP) control in patients with uncontrolled hypertension (HTN). The work builds on our experience in implementing new models of care in Veterans Affairs (VA) and non-VA settings, including three National Institute of Health (NIH) studies of pharmacist-based HTN management. The long-term effectiveness of such models, especially in veterans, is unknown. Thus, the primary goal of this study is to evaluate how to sustain long-term BP control in veterans with HTN following a 6-month intensive pharmacist intervention.

This study will enroll veterans with uncontrolled HTN into a 6-month intensive pharmacist-based intervention. Following this initial intervention, participants will be randomized to continued intervention or a one-time patient and provider education intervention. BP will be compared in the two groups over a 2-year follow-up period. The intervention to control and sustain BP will follow VA guidelines and include: 1) comprehensive medication assessment by the pharmacist; 2) an explicit plan to intensify treatment if indicated; 3) strategies to improve adherence; and 4) follow-up pharmacist visits to sustain BP control. The intervention is based on models identified in a recent Agency for Healthcare Research and Quality (AHRQ) report as being the most potent strategies to improve BP. The study will benefit from a strong research team with expertise in guideline development, implementation science, quality measurement, and behavioral science. The study will also provide important information on the degree to which BP control deteriorates after patients are referred back to usual care. The specific aims and related hypotheses of the study are to:

Aim 1:Compare BP control in patients randomized to long-term continuation of the pharmacist intervention or to a less intense one-time patient and provider education intervention.

Hypothesis 1a: Patients randomized to the continued pharmacist intervention will have higher rates of BP control 24 months after randomization.

Hypothesis 1b: Patients randomized to the continued pharmacist intervention will have lower mean BP 24 months after randomization.

Aim 2: Compare antihypertensive medication intensification in patients randomized to the continued pharmacist intervention or the less intense intervention.

Hypothesis 2: A higher proportion of patients who continued the pharmacist intervention will have medication intensification over the 24-month follow-up.

Aim 3: Compare medication adherence in the two intervention groups. Hypothesis 3a: Medication adherence will be higher in patients randomized to the continued pharmacist intervention group during the 24 month follow-up period.

Hypothesis 3b: Improvements in medication adherence will be associated with improvements in BP during each study interval.

DETAILED DESCRIPTION:
We are proposing a 4-year trial to determine if long-term blood pressure (BP) control after a pharmacist intervention requires continuation of the intervention or if a less intense strategy is equally efficacious. The intervention builds on the Chronic Care Model, recent Veteran Affairs (VA) trials, and our pharmacist interventions. This research has convincingly shown that collaborative interventions can improve BP control over 6-9 months. However, no randomized study has evaluated strategies to sustain the effect of such interventions.

The study will enroll 300 patients with uncontrolled HTN at the Iowa City Veteran Affairs Medical Center (VAMC) and an affiliated community based outpatient clinic (CBOC). All patients will receive a pharmacist intervention for 6 months that will follow VA HTN guidelines. Patients completing the intervention will then be randomized to continuation of the high intensity intervention or to a one-time patient and provider education intervention that was recently shown to be effective. The high intensity (HI) intervention will intensify medication regimens when BP deteriorates, sustain adherence, and improve monitoring to reduce adverse drug reactions. The low intensity (LI) intervention will involve usual care by patients primary care provider (PCPs) and a one-time education intervention including a letter emphasizing the importance of medication adherence and behavioral strategies to improve BP control (e.g., low-salt diets, exercise). PCPs of low intensity patients will also receive a computerized alert with treatment recommendations and links to BP guidelines.

The primary endpoint-BP-will be assessed using standard measurements at 6, 12, 18, 24, and 30 months post enrollment (24 months after randomization). The 24-month evaluation phase will determine if BP control can be sustained or improved with a continued high intensity intervention, relative to a low intensity intervention (Aim 1). All medication changes will be assessed to compare rates of medication intensification over the follow-up period (Aim 2). Finally, validated self-report adherence questionnaires will be used to compare medication adherence in the two groups and determine relationships between BP control and medication adherence (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hypertension (HTN) captured by ICD-9-CM codes from prior outpatient visits;
* elevated BP (>140/90 mmHg among non-diabetics; or >140/80 mmHg among diabetics) during the most recent VA clinic visit or based on the average from the last 3 visits;
* elevated BP measured by the Research Medical Assistant (MA) at the baseline visit.

Exclusion Criteria:

Patients will be excluded for the following safety reasons:

* prior history or current signs of hypertensive emergency including symptoms of angina, stroke, or acute renal failure;
* severe HTN (systolic BP >200 or diastolic BP > 114mm Hg);
* history of acute MI, stroke, or unstable angina in the prior 6 months;
* Congestive Heart Failure (CHF) due to systolic dysfunction with a left ventricular ejection fraction < 35% documented by echocardiography, nuclear medicine study, or ventriculography;
* renal insufficiency, defined by a glomerular filtration rate less than 30 ml/min or previously documented proteinuria > 1 gram per day;
* significant hepatic disease, including prior diagnoses of cirrhosis, Hepatitis B or C infection, or laboratory abnormalities (serum ALT or AST > 2 times control or total bilirubin > 1.5 mg/dl) in the prior 6 months;
* pregnancy;
* prior diagnoses of pulmonary hypertension or sleep apnea (unless treated by continuous positive pressure ventilation);
* poor prognosis with a life expectancy estimated less than 2 years;
* residence in a nursing home or diagnosis of dementia;
* inability to give informed consent or impaired cognitive function (defined as > 3 errors on the 10-item Pfeiffer Portable Mental Status Questionnaire, administered during study intake);
* no telephone for follow-up calls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E. Rosenthal, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

REFERENCES:
- [Result] Carter BL, Coffey CS, Uribe L, James PA, Egan BM, Ardery G, Chrischilles EA, Ecklund D, Vander Weg M, Vaughn T; Collaboration Among Pharmacists and Physicians to Improve Outcomes Now (CAPTION) trial investigators. Similar blood pressure values across racial and economic groups: baseline data from a group randomized clinical trial. J Clin Hypertens (Greenwich). 2013 Jun;15(6):404-12. doi: 10.1111/jch.12091. Epub 2013 Apr 1. PMID 23730989
- [Result] Parker CP, Cunningham CL, Carter BL, Vander Weg MW, Richardson KK, Rosenthal GE. A mixed-method approach to evaluate a pharmacist intervention for veterans with hypertension. J Clin Hypertens (Greenwich). 2014 Feb;16(2):133-40. doi: 10.1111/jch.12250. PMID 24588813
- [Result] Carter BL, Chrischilles EA, Rosenthal G, Gryzlak BM, Eisenstein EL, Vander Weg MW. Efficacy and safety of nighttime dosing of antihypertensives: review of the literature and design of a pragmatic clinical trial. J Clin Hypertens (Greenwich). 2014 Feb;16(2):115-21. doi: 10.1111/jch.12238. Epub 2013 Dec 24. PMID 24373519
- [Result] Hawkins MS, Hough LJ, Berger MA, Mor MK, Steenkiste AR, Gao S, Stone RA, Burkitt KH, Marcus BH, Ciccolo JT, Kriska AM, Klinvex DT, Sevick MA. Recruitment of veterans from primary care into a physical activity randomized controlled trial: the experience of the VA-STRIDE study. Trials. 2014 Jan 7;15:11. doi: 10.1186/1745-6215-15-11. PMID 24398076
- [Derived] Carter BL, Vander Weg MW, Parker CP, Goedken CC, Richardson KK, Rosenthal GE. Sustained Blood Pressure Control Following Discontinuation of a Pharmacist Intervention for Veterans. J Clin Hypertens (Greenwich). 2015 Sep;17(9):701-8. doi: 10.1111/jch.12577. Epub 2015 Jun 1. PMID 26032843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 249 total were enrolled. 122 had controlled BP and did not participate in the trial. of the 127 who participated, 4 dropped prior to randomization.
Groups:
- Arm 2: VA patients with uncontrolled HTN.
  Low Intensity Intervention: Patients randomized to the low intensity group will receive management by their PCP and a three-part intervention that was effective in a recent VA study.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 61 | 62
Completed | 48 | 52
Not Completed | 13 | 10
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (11.2) | 66.0 (10.3) | 64.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 60 | 60 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 57 | 57 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 61 | 62 | 123

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Change
Description: Participant's Blood Pressure (BP) will be measured using a standard protocol following American Heart Association guidelines using an Omron HEM 907 device. The primary endpoint-BP-will be assessed using standard measurements at baseline, 6, 12, 18, 24, and 30 months post enrollment (24 months after randomization).
Time Frame: Measured at Baseline, and 6,12,18,24, and 30 months post baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 48 | 52
mmHg
  Basline Systolic BP | 148 (14) | 147 (12)
  Baseline Diastolic BP | 79 (11) | 79 (10)
  6-month Systolic BP | 134 (16) | 135 (14)
  6-month Diastolic BP | 73 (12) | 74 (10)
  12-month Systolic BP | 136 (17) | 135 (16)
  12-month Diastolic BP | 75 (11) | 74 (10)
  18-month Systolic BP | 135 (17) | 137 (18)
  18-month Diastolic BP | 73 (9) | 75 (10)
  24-month Systolic BP | 134 (17) | 135 (16)
  24-month Diastolic BP | 73 (9) | 74 (9)
  30-month Systolic BP | 131 (17) | 136 (17)
  30-month Diastolic BP | 72 (11) | 73 (11)

ADVERSE EVENTS:
Description: All study participants are counted in the Number of Participants at Risk. No Other Adverse Events were observed.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/62
Other Adverse Events (participants affected / at risk) | 0/61 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=61) | Arm 2 (N=62)
Drug--Participant Hospitalization (General disorders) | 1 (1) | 0 (0) — The participant was admitted to a medicine unit for workup of his hyponatremia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes